CLINICAL TRIAL: NCT05358184
Title: High Frequency Percussive Ventilation in COVID-19 Patients Receiving Oxygen Through High-flow Nasal Cannula
Brief Title: High Frequency Percussive Ventilation in COVID-19 Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Magna Graecia (Other)
Responsible Party: Principal Investigator, Federico Longhini, Director of the Intensive Care and Anesthesia Department, University Magna Graecia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Percussionaire COVID
Record Dates: First submitted 2022-04-29; First posted 2022-05-03 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: COVID-19; Acute Respiratory Failure
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High frequency percussive ventilation (Experimental): High Frequency Percussive Ventilation will be applied for 10 minutes at an oscillation frequency of 10 Hz, superimposed to oxygen therapy at high flow through nasal cannula
  Interventions: Device: High frequency Percussive ventilation

INTERVENTIONS:
Device: High frequency Percussive ventilation — High Frequency Percussive Ventilation will be applied for 10 minutes at an oscillation frequency of 10 Hz

SUMMARY:
High frequency percussive ventilation (HFPV) is used in patients with underlying pulmonary atelectasis, excessive airway secretions, and respiratory failure. HFPV is a non-continuous form of high-frequency ventilation delivered by a pneumatic device that provides small bursts of sub-physiological tidal breaths at a frequency of 60-600 cycles/minute superimposed on a patient's breathing cycle. The high-frequency breaths create shear forces causing dislodgement of the airway secretions. Furthermore, the HFPV breath cycle has an asymmetrical flow pattern characterized by larger expiratory flow rates, which may propel the airway secretions towards the central airway. In addition, the applied positive pressure recruits the lung units, resulting in a more homogeneous distribution of ventilation and improved gas exchange. In acute care and critical care settings, HFPV intervention is used in a range of patients, from spontaneously breathing patients to those receiving invasive mechanical ventilation where HFPV breaths can be superimposed on a patient's breathing cycle or superimposed on breaths delivered by a mechanical ventilator. The most common indications for HFPV use are reported as removal of excessive bronchial secretions, improving gas exchange, and recruitment of atelectatic lung segments. This study aims to assess the lung physiological response to HFPV in terms of aeration and ventilation distribution in patients with acute respiratory failure due to SARS-CoV-2 infection and requiring high flow oxygen therapy through nasal cannula

ELIGIBILITY:
Inclusion Criteria:

* acute respiratory failure with a nasal swab positive for SARS-CoV-2
* need for high-flow oxygen through nasal cannula

Exclusion Criteria:

* life threatening cardiac arrythmia
* pneumothorax
* acute spinal injury
* chest trauma
* hemodynamic instability
* chest or abdominal surgery in the previous 7 days
* pregnancy
* enrollment in other study protocols

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-05-15 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Lung aeration | 5 minutes after the end of HFPV application
  To evaluate if the application of High Frequency Percussive Ventilation (HFPV) will modify the lung aeration (as assessed by the end-expiratory lung impedance through EIT), as compared to baseline before the treatment
Lung aeration | One hour after the end of HFPV application
  To evaluate if the application of High Frequency Percussive Ventilation (HFPV) will modify the lung aeration (as assessed by the end-expiratory lung impedance through EIT), as compared to baseline before the treatment
Lung aeration | Three hours after the end of HFPV application
  To evaluate if the application of High Frequency Percussive Ventilation (HFPV) will modify the lung aeration (as assessed by the end-expiratory lung impedance through EIT), as compared to baseline before the treatment

SECONDARY OUTCOMES:
Gas exchange | 5 minutes after the end of HFPV application
  To evaluate if the application of High Frequency Percussive Ventilation (HFPV) will modify Arterial Blood Gases, as compared to baseline before the treatment
Gas exchange | One hour after the end of HFPV application
  To evaluate if the application of High Frequency Percussive Ventilation (HFPV) will modify Arterial Blood Gases, as compared to baseline before the treatment
Gas exchange | Three hours after the end of HFPV application
  To evaluate if the application of High Frequency Percussive Ventilation (HFPV) will modify Arterial Blood Gases, as compared to baseline before the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Federico Longhini, MD, Principal Investigator — Magna Graecia University

IPD SHARING:
Plan to Share IPD: Yes
Anonymous data will be shared after study publication on a peer-reviewed journal in english language, on a reasonable request to the principal investigator
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: After study publication on a peer-reviewed journal in english language
Access Criteria: On reasonable request to the Principal Investigator